CLINICAL TRIAL: NCT03912727
Title: A Protective Role of Alpha Lipoic Acid Against Possible Cardiovascular Events in Patients With Haemodialysis
Brief Title: Alpha Lipoic Acid Against Cardiovascular Events in Patients With Haemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehab Werida (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor-Investigator, Rehab Werida, Lecturer, Damanhour University
Organization: Damanhour University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ALA in haemodialysis
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Hemodialysis Complication
Keywords: alpha-lipoic acid; Cardiovascular events; Hemodialysis
MeSH Terms: interventions — Thioctic Acid; Renal Replacement Therapy

STUDY DESIGN:
Intervention Model Description: 36 patients with end-stage renal disease (ESRD) receiving hemodialysis treatment will be enrolled in the study and the patients will be identified by coded numbers to maintain the privacy.
  Patients will be randomized into two groups each group includes 18 patients:
  Control Group: 18 patients will receive their standard therapy only. Tested Group: 18 patients will receive alpha lipoic acid (thiotacidR) product with their standard therapy.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpha-lipoic acid (Experimental): 18 patients will receive alpha lipoic acid (thiotacidR) product with their standard therapy.
  Interventions: Dietary Supplement: Alpha-Lipoic acid plus renal replacement therapy; Other: renal replacement therapy
- Control (Placebo Comparator): 18 patients will receive their standard therapy only.
  Interventions: Other: renal replacement therapy

INTERVENTIONS:
Dietary Supplement: Alpha-Lipoic acid plus renal replacement therapy — Alpha lipoic acid (ALA) is a vitamin-like antioxidant
  Other Names: Thiotacid ( Alpha-Lipoic acid 600 mg )
  Arms: Alpha-lipoic acid
Other: renal replacement therapy — standard renal replacement therapy

SUMMARY:
Evaluate the association between possible benefit effects of oral administration of alpha lipoic acid by patients with hemodialysis and the possible reduction in cardiovascular events (CVEs); using Advanced glycation end products (AGEs) as a measure to assess endothelium function which correlate with CVEs.

DETAILED DESCRIPTION:
Study design: double blind, Parallel, Randomized, Prospective, Controlled study. Setting: Nephrology Department, Dialysis units, Ain Shams University Hospitals, Ain Shams University, Cairo, Egypt.

Sample size:

36 patients with end-stage renal disease (ESRD) receiving dialysis treatment will be enrolled in the study and the patients will be identified by coded numbers to maintain the privacy.

Patients will be randomized into two groups each group includes 18 patients:

Control Group: 18 patients will receive their standard therapy only. Tested Group: 18 patients will receive alpha-lipoic acid (thiotacid R) product with their standard therapy.

Materials:

Thiotacid R 600 mg tablet. Each tablet contains: Thioctic acid (Alpha-lipoic acid) 600 mg; a product of EVA pharma, Cairo, Egypt.

Methods:

All Patients will be subjected to the following:

1. Informed consent
2. Demographics and history taking: Using Patient Data sheet
3. Laboratory evaluation including:

   A- Routine laboratory measurements as hemoglobin, calcium, phosphate, and albumin will be determined.

   The assessment will be done in 2 occasions:

   i. At Baseline (before the beginning of the treatment) for all groups ii. After 3 months of addition of alpha lipoic acid to their standard therapy for the tested group.
4. Follow up:

A- During-treatment follows up of the patients:

All patients will be followed up during the study for treatment tolerability by assessing adverse effects, and compliance to drug regimen.

Drug regimen: - the patients in tested group will administered Thiotacid 600 mg; orally once daily for 3 months as add on the standard therapy that are receiving.

Patients will be interviewed weekly through face to face contact with the clinical pharmacist regarding treatment tolerability, and through telephone calls in between these weekly meetings.

B- Post-treatment follows up of the patients:

All patients in control group will be followed up clinically after 3 months from the start of the study and all laboratory examinations will be carried out.

All patients in tested group will be followed up clinically after 3 months from the start of treatment and all laboratory examinations will be carried out.

ELIGIBILITY:
IPatients eligible for the study fulfilled the following inclusion criteria and free from exclusion criteria:

Inclusion criteria:

1. Clinical stable patients on hemodialysis for at least 3 months.
2. Aged between18 - 60 years old.
3. Both sexes.
4. Patients who accept to participate in the study.

Exclusion criteria:

1. The patients suffering from other diseases, which may lead to oxidative stress, such as: Inflammatory diseases, hepatic or respiratory diseases …
2. Smokers and alcoholics
3. Non-compliant patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Advanced glycation and oxidation end products (AGEs) | three months
  Blood AGEs concentration was measured by fluorescence emission

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab A Zalat, Ass. Prof., Study Director — Al-Azhar University
Locations (1):
- Nephrology Department, Dialysis units, Ain Shams University Hospitals, Ain Shams University, Cairo, Egypt., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rivara MB, Yeung CK, Robinson-Cohen C, Phillips BR, Ruzinski J, Rock D, Linke L, Shen DD, Ikizler TA, Himmelfarb J. Effect of Coenzyme Q10 on Biomarkers of Oxidative Stress and Cardiac Function in Hemodialysis Patients: The CoQ10 Biomarker Trial. Am J Kidney Dis. 2017 Mar;69(3):389-399. doi: 10.1053/j.ajkd.2016.08.041. Epub 2016 Dec 4. PMID 27927588
- [Background] Liakopoulos V, Roumeliotis S, Bozikas A, Eleftheriadis T, Dounousi E. Antioxidant Supplementation in Renal Replacement Therapy Patients: Is There Evidence? Oxid Med Cell Longev. 2019 Jan 15;2019:9109473. doi: 10.1155/2019/9109473. eCollection 2019. PMID 30774749